CLINICAL TRIAL: NCT00006017
Title: A Randomized Phase II Trial of Two Different Schedules of Administration of Rebeccamycin Analog in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Two Rebeccamycin Analogue Regimens in Treating Patients With Advanced or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Afshin Dowlati, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1599; U01CA063200 (NIH); P30CA043703 (NIH); CWRU-1599; NCI-91
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — becatecarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rebeccamycin 1 day (Active Comparator): Patients receive rebeccamycin analogue IV over 1 hour on day 1.
  Interventions: Drug: becatecarin
- Rebeccamycin 5 day (Active Comparator): Patients receive rebeccamycin analogue IV over 1 hour on days 1-5.
  Interventions: Drug: becatecarin

INTERVENTIONS:
Drug: becatecarin — Arm I: Patients receive rebeccamycin analogue IV over 1 hour on day 1. Arm II: Patients receive rebeccamycin analogue IV over 1 hour on days 1-5. Treatment for both arms repeats every 3 weeks for 6-8 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: DEAE-rebeccamycin; rebeccamycin analogue; rebeccamycin analogue, tartrate salt

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of rebeccamycin analogue is more effective in treating non-small cell lung cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of two rebeccamycin analogue regimens in treating patients who have stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy, in terms of response rate, in patients with advanced or recurrent non-small cell lung cancer treated with rebeccamycin analogue via 1 infusion vs 5 daily infusions every 3 weeks.
* Compare the response duration in patients treated with these regimens.
* Compare the toxicity profiles of these two regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to performance status (0 or 1 vs 2) and participating center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive rebeccamycin analogue IV over 1 hour on day 1.
* Arm II: Patients receive rebeccamycin analogue IV over 1 hour on days 1-5. Treatment for both arms repeats every 3 weeks for 6-8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 36-64 patients (18-32 per arm) will be accrued for this study at a rate of 3-4 patients per month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IIIB (with pleural effusions), IV, or recurrent non-small cell lung cancer with failure on 1 prior chemotherapy regimen
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT less than 2 times normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 1 prior chemotherapy regimen
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent combination antiretroviral therapy for HIV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2000-05; Primary Completion 2003-07 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy, in terms of response rate, in patients with advanced or recurrent non-small cell lung cancer treated with rebeccamycin analogue | via 1 infusion vs 5 daily infusions every 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio